CLINICAL TRIAL: NCT04077177
Title: Decreasing Body Dissatisfaction in Male College Athletes: A Randomized Controlled Trial of the Male Athlete Body Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Institute of Technology (Other)
Collaborators: DePaul University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IllinoisIT
Record Dates: First submitted 2019-08-05; First posted 2019-09-04 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment Only (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Male Athlete Body Project

INTERVENTIONS:
Behavioral: Male Athlete Body Project — Participants who meet eligibility criteria and consent to the study will be randomized to one of two conditions: intervention condition (i.e., Male Athlete Body Project) or an assessment only control condition. The intervention groups will take place at IIT. Participants who accept randomization to condition will complete baseline questionnaires after randomization (immediately prior to Session 1 in the intervention condition and after being randomized to the assessment only control condition). Questionnaires will be repeated immediately post-intervention (intervention condition)/after a 3-week interval (control). All participants will be asked to complete the questionnaires again, 4 weeks after the previous round of questionnaires. The 3, 80-minute group sessions will be separated by 1 week.
  Arms: Intervention

SUMMARY:
Body Dissatisfaction (BD) is associated with marked distress and often precipitates disordered eating symptomology (Milligan & Pritchard, 2006). BD in male athletes is an important area to explore, as research in this field often focuses on eating disorders in female athletes (e.g., Becker et al., 2012; Varnes et al., 2013). The current body of literature regarding male college athletes suggests that they experience pressures associated with both societal muscular ideals and sport performance (Galli et al., 2015). While there is a clear association between drive for muscularity and BD in collegiate male athletes (Galli et al., 2015), no study to date has conducted research aimed to attenuate the effect of BD in this population. The current study seeks to investigate a BD intervention for male college athletes. Participants will be randomized to an adapted version of the standardized Female Athlete Body Project (i.e., the Male Athlete Body Project) or an assessment only control condition. All participants will complete baseline and post-treatment measures of BD, negative affect, internalization of an athletic ideal, drive for muscularity, sport confidence, eating pathology, and unhealthy weight-control behaviors. Study aims are to determine if the Male Athlete Body Project intervention group reduces BD and related factors post-treatment, and to investigate whether these differences are maintained at 1-month follow up. Results will inform mental health and sport clinicians, coaches, and other personnel involved in an athlete's care about successful strategies for decreasing BD.

ELIGIBILITY:
Inclusion Criteria:

* Male
* member of a university-sponsored varsity athletic team
* over age 18
* some endorsement of body dissatisfaction (i.e., scores greater than zero). To maximize generalizability, there are no additional inclusion criteria, consistent with recommendations from previous athlete Body Project research

Exclusion Criteria:

* NONE

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 83 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change is being assessed with Multidimensional Body-Self Relations Questionnaire (MBSRQ) - Appearance Scale | Participants will complete this at baseline, 3-week follow up, and 1-month follow-up
  This measure assesses body dissatisfaction and appearance concerns over 34 items. The total score will not be interpreted; instead, subscale scores will be reported and interpreted. The subscales are: Appearance Evaluation, Appearance Orientation, Overweight Preoccupation, Self-Classified Weight, and the Body Areas Satisfaction Scale. For the Appearance Evaluation subscale, higher scores indicate a better outcome. Scores range from 7-35. For Appearance Orientation, higher scores indicate a worse outcome. Scores range from 12-60. For the Overweight Preoccupation subscale, higher scores represent a worse outcome. Scores range from 4-20. For Self-Classified Weight, higher scores represent the individual believing they are overweight. Scores range from 2-8. For the Body Areas Satisfaction Scale, higher scores indicate a better outcome. Scores range from 9-45.

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perelman H, Schwartz N, Yeoward-Dodson J, Quinones IC, Murray MF, Dougherty EN, Townsel R, Arthur-Cameselle J, Haedt-Matt AA. Reducing eating disorder risk among male athletes: A randomized controlled trial investigating the male athlete body project. Int J Eat Disord. 2022 Feb;55(2):193-206. doi: 10.1002/eat.23665. Epub 2022 Jan 17. PMID 35037275